CLINICAL TRIAL: NCT03362996
Title: Randomized, Double Blind, Placebo Controlled Prospective Study, to Evaluate the Effect of Freshly-Pressed Extra Virgin Olive Oil in the Disease's Progression in Patients Diagnosed With Mild Cognitive Impairment
Brief Title: Management of Mild Cognitive Impairment Patients With Extra Virgin Olive Oil - MICOIL
Acronym: MICOIL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Greek Alzheimer's Association and Related Disorders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25/201614
Record Dates: First submitted 2017-11-03; First posted 2017-12-05 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Mild Cognitive Impairment
Keywords: extra virgin olive oil; mild cognitive impairment; randomized double blind clinical trial
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (Experimental): 50 patients Freshly-Pressed Extra Virgin Olive Oil Aluminum bottle with 500 ml of freshly-pressed extra virgin olive oil 1 bottle per 10 days.
  Dietary Supplement: Freshly-Pressed Extra Virgin Olive Oil dietary intake of the content of 50 mL (3 tablespoons from the bottle containing the product)
  Interventions: Dietary Supplement: Freshly-Pressed Extra Virgin Olive Oil
- Control group 1 (Placebo Comparator): 50 patients Extra Virgin Olive Oil Aluminum bottle with 500 ml of freshly-pressed extra virgin olive oil 1 bottle per 10 days. Extra Virgin Olive Oil dietary intake of the content of 50 mL (3 tablespoons from the bottle containing the product)
  Interventions: Combination Product: extra virgin olive oil
- Control Group 2 (Other): 50 patients that will have the same dietary habits and a Mediterranean dietary protocol
  Interventions: Other: mediterranean diet

INTERVENTIONS:
Dietary Supplement: Freshly-Pressed Extra Virgin Olive Oil — Dietary Supplement: Freshly-pressed extra virgin olive oil Freshly-Pressed Extra Virgin Olive Oil Aluminum bottle with 500 ml of freshly-pressed extra virgin olive oil 1 bottle per 10 days
  Arms: Experimental Group
Combination Product: extra virgin olive oil — Extra Virgin Olive Oil Aluminum bottle with 500 ml of freshly-pressed extra virgin olive oil 1 bottle per 10 days
  Arms: Control group 1
Other: mediterranean diet — 50 patients that will have the same dietary habits and a Mediterranean dietary protocol
  Arms: Control Group 2

SUMMARY:
There is accumulating evidence suggesting that olive oil may have a positive impact on conditions involving cognitive deficits, such as MCI and AD. More specifically, these beneficial effects are mostly attributed to some phenolic compounds in olive oil, such as oleocanthal, oleuropein and ligstroside. Oleocanthal is deeper studied than the rest of olive oil phenol components and it shows promising results in neuroprotection against AD through various suggested mechanisms, such as the enhancement of amyloid-beta clearance in the brain and the inhibition of neurofibrillary tangles formation. For this reason, it would be interesting to study the effects of freshly-pressed extra virgin olive oil, as it is known that it contains oleocanthal in higher concentrations than the normal extra virgin olive oil. The aim of the study is to evaluate the beneficial effect of extra virgin olive oil in comparison to freshly-pressed extra virgin olive oil on patients diagnosed with mild cognitive impairment (MCI).

Study Type: Interventional Study Design: Allocation: Randomized Intervention Model: Parallel Assignment Masking: Double Blind (Subject, Investigator) Primary Purpose: Prevention

DETAILED DESCRIPTION:
OBJECTIVES OF THE TRIAL

The objectives of this study are:

* To investigate the efficacy of freshly pressed EVOO as a disease course modifying treatment for mild cognitive impairment in a phase III double-blind placebo-controlled study.
* To investigate the effects in objective measurements in patients with mild cognitive impairment.

STUDY DESIGN This is a Greek, randomized, double-blind, placebo-controlled study group of EVOO compared with placebo. Qualifying patients will be randomly assigned to receive 50mL of freshly-pressed EVOO or placebo (EVOO) or mediterranean dietary protocol on a daily basis for 24 months. Patients undergo assessments at baseline,12 and 24 months +/- 7 days after beginning treatment.

Duration The total study duration will be 30 months. Patients will receive study medication for 24 months.

Number of Subjects 150 subjects total will be enrolled. ; 50 in the experimental group (freshly pressed EVOO); 50 in the Control Group 1(EVOO) and 50 in control Group 2(same dietary habits-mediterranean dietary protocol).

Patient Eligibility Screening Form (ESF)

An eligibility form documenting the patient's fulfillment of the entry criteria will be completed by the assessor. The following information will be included in the ESF:

* Patient identification: Initials (First initial of first name and First initial of surname), date of birth and Patient Identification Number.
* Eligibility Screening; Checklist of inclusion and exclusion criteria
* Eligibility Statement; for patients found to be ineligible, the reason for ineligibility must be stated
* Written informed consent will be obtained from the subject . The informed consent form must be co-signed by the physician. The nature of the study and the potential risks associated with the trial will be explained to all subject candidates and their responsible informants.
* Signature and date: the ESF may be completed by an assessor but it is required that the principal investigator/study clinician sign and date the ESF to verify eligibility of the patient for inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Memory Complaints
* Abnormal memory function documented by scoring 1 SD below the age-adjusted mean on the Logical Memory II subscale, (Delayed Paragraph Recall) from the Wechsler Memory Scale-R.
* MMSE 24-30
* CDR(sum of boxes) >= 0,5
* Diagnosis: Mild Cognitive Impairment (amnestic plus multi-domain)
* Geriatric Depression Scale (GDS) <6
* Hachinski Modified Ischemic scale <= 4
* Stability of Permitted Medications for 4 weeks
* Years of education: >= 5
* Proficient language fluency
* Have a study partner with 10+ hr/wk contact (can be in person and telephone), accompanies to visits
* Compliance

Exclusion Criteria:

* Visual and auditory acuity inadequate for neuropsychological testing
* Enrollment in other trials or studies not compatible with MICOIL
* History of significant neurological or psychiatric illnesses or presence of other diseases precluding enrollment.
* Use of forbidden medications (listed below)
* Ferromagnetic implants and devices (including implants or devices held in place by sutures, granulation or ingrowth of tissue, fixation devices, or by other means) not eligible for MRI scanning. Brain malformation or other conditions that may complicate lumbar puncture

Medications across the study

Excluded Medication:

* Antidepressants with anti-cholinergic properties.
* Regular use of narcotic analgesics (>2 doses per week) within 4 weeks of screening.
* Use of neuroleptics with anti-cholinergic properties (e.g., chlorpromazine, thioridazine) within 4 weeks of screening.
* Chronic use of other medications with significant central nervous system anticholinergic activity within 4 weeks of screening (e.g., diphenhydramine).
* Use of Anti-Parkinsonian medications (including Sinemet, amantadine, bromocriptine, pergolide, selegeline) within 4 weeks of screening.
* Participation in any other investigational drug study within 4 weeks of screening (individuals may not participate in any drug study while participating in this protocol).

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-11-09 (Actual); Primary Completion 2018-02-15 (Estimated); Study Completion 2019-05-15 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological Assessment- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in Mini-Mental State Examination (MMSE) score
FUCAS-Measurements to Assess Daily Functionality | baseline, 12 and 24 months
  Changes in Functional cognitive assessment scale (FUCAS) score
Letter & Category Fluency Test- Measurement to Assess Verbal Fluency and Learning | baseline, 12 and 24 months
  Changes in the Letter & Category Fluency Test
CDR- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in Global Clinical Dementia Rating (CDR) score (sum of boxes)
MoCA- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in Montreal Cognitive Assessment (MoCA)
CANTAB- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in Cambridge Neuropsychological Test Automated Battery (CANTAB)
Clock Drawing test- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in the Clock Drawing test
Logical Memory test- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in the Logical Memory test
Digit Span Forward & Backward test- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in the Digit Span Forward & Backward test
WAIS-R Digit Symbol- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in the WAIS-R Digit Symbol Substitution Test
TMT part A and B- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in the Trail Making Test
ADASCog-Measurements to Assess Daily Functionality | baseline, 12 and 24 months
  Changes in Alzheimer's Disease Assessment Scale-Cognitive (ADASCog)
Functional Rating Scale for Dementia-Measurements to Assess Daily Functionality | baseline, 12 and 24 months
  Changes in Functional Rating Scale for Dementia (FRSSD)
Auditory Verbal Learning Test- Measurement to Assess Verbal Fluency and Learning | baseline, 12 and 24 months
  Changes in the Auditory Verbal Learning Test
Boston Naming Test- Measurement to Assess Verbal Fluency and Learning | baseline, 12 and 24 months
  Changes in the Boston Naming Test

SECONDARY OUTCOMES:
NeuroImaging | baseline and 24 months
  Changes in brain Magnetic Resonance Imaging (MRI) 1.5 Tesla (brain atrophy) [Time Frame: baseline, 24 month]
CSF - beta amyloid | baseline and 24 months
  Changes in mean values on high sensitivity beta-amyloid 1-42 protein
CSF TAU-protein | baseline and 24 months
  Changes in mean values on TAU-protein in cerebrospinal fluid
Neurophysiology and ERPs | baseline, 12 and 24 months
  •Changes in Event-Related Potential (ERP) (oddball paradigm, auditory ERPs) [Time frame: baseline, 12 month, 24 month]
Electroencephalography recording | baseline, 12 and 24 months
  •Changes in Electroencephalography (EEG), resting state.The device records brain signals through 57 electrodes, 2 reference electrodes attached to the earlobes, and a ground electrode placed at a left anterior position. [Time frame: baseline, 12 month, 24 month]

OTHER OUTCOMES:
Weight in Kilograms | baseline, 12 and 24 months
  Changes in weight
Height in Meters | baseline, 12 month and 24 month
  Changes in Height

CONTACTS AND LOCATIONS:
Overall Officials: Magda Tsolaki, Professor, Principal Investigator — Greek Alzheimer's Association and Related Disorders
Locations (1):
- Greek Association of Alzheimer's Disease and Related Disordeers, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided
Not available at this stage

REFERENCES:
- [Background] Tsolaki M, Karathanasi E, Lazarou I, Dovas K, Verykouki E, Karacostas A, Georgiadis K, Tsolaki A, Adam K, Kompatsiaris I, Sinakos Z. Efficacy and Safety of Crocus sativus L. in Patients with Mild Cognitive Impairment: One Year Single-Blind Randomized, with Parallel Groups, Clinical Trial. J Alzheimers Dis. 2016 Jul 27;54(1):129-33. doi: 10.3233/JAD-160304. PMID 27472878
- [Derived] Tzekaki EE, Tsolaki M, Geromichalos GD, Pantazaki AlphaA. Extra Virgin Olive Oil consumption from Mild Cognitive Impairment patients attenuates oxidative and nitrative stress reflecting on the reduction of the PARP levels and DNA damage. Exp Gerontol. 2021 Dec;156:111621. doi: 10.1016/j.exger.2021.111621. Epub 2021 Nov 5. PMID 34748951
- [Derived] Tzekaki EE, Tsolaki M, Pantazaki AlphaA, Geromichalos G, Lazarou E, Kozori M, Sinakos Z. The pleiotropic beneficial intervention of olive oil intake on the Alzheimer's disease onset via fibrinolytic system. Exp Gerontol. 2021 Jul 15;150:111344. doi: 10.1016/j.exger.2021.111344. Epub 2021 Apr 6. PMID 33836262